CLINICAL TRIAL: NCT07108010
Title: Evaluation of ABO and Rh Blood Group Frequencies in Acute Leukemia
Brief Title: ABO and Rh Blood Group Frequencies in Acute Leukemia Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aisha Abobakr Abass Metwally, Clinical Pathology Resident / M.Sc. Candidate, South Egypt Cancer Institute, Assiut University, Assiut University
Other Study IDs: Blood group in Acute Leukemia
Record Dates: First submitted 2025-07-31; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Acute Leukemia (Including Acute Myeloid Leukemia and Acute Lymphoblastic Leukemia)
Keywords: Acute Leukemia; ABO Blood Group and Rh Blood Group; Hematologic Malignancies; Retrospective Study
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective observational study aims to evaluate the distribution of ABO and Rh blood groups among patients diagnosed with acute leukemia. By analyzing medical records from leukemia cases, the study seeks to identify any potential associations between blood group types and the occurrence of the disease.

DETAILED DESCRIPTION:
Acute leukemia is a group of hematologic malignancies characterized by the rapid proliferation of immature blood cells, leading to bone marrow failure and systemic complications. It is broadly classified into two main types: acute lymphoblastic leukemia (ALL) and acute myeloid leukemia (AML), depending on the lineage of the malignant cells. Despite advancements in the understanding of leukemia pathogenesis, the etiology remains multifactorial and incompletely understood.

Recent studies have suggested a potential association between blood group antigens-particularly those of the ABO and Rh systems-and the risk of developing various types of cancer, including hematological malignancies. The ABO antigens are expressed not only on red blood cells but also on epithelial and endothelial cells, and may influence cancer biology through mechanisms involving immune response modulation, cell adhesion, and inflammation.

Several epidemiological investigations have explored the relationship between ABO and Rh blood groups and malignancies such as gastric, pancreatic, breast, and hematologic cancers. However, data regarding their association with acute leukemia are still limited, inconsistent, and often vary across different populations and study designs.

This study is a retrospective observational analysis conducted at the Clinical Pathology Department, South Egypt Cancer Institute, Assiut University. It aims to assess the frequencies of ABO and Rh blood groups among patients diagnosed with acute leukemia over a defined period. The findings will be compared to blood group distributions in healthy blood donors to explore any statistically significant associations.

Understanding whether certain blood group antigens are associated with an increased or decreased risk of acute leukemia may help identify at-risk individuals, contribute to risk stratification, and provide further insight into the biology of leukemogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with de-novo acute leukemia (ALL or AML)
* Diagnosis confirmed between 2022 and 2025
* ABO and Rh blood group data available
* Patients treated at or referred to South Egypt Cancer Institute, Assiut University

Exclusion Criteria:

* Incomplete or missing blood group data
* Presence of other malignancies or chronic systemic illnesses
* History of blood transfusion prior to diagnosis or blood grouping

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with de-novo acute leukemia (ALL and AML) at South Egypt Cancer Institute, Assiut University, during the period from 2022 to 2025.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-04-28 (Estimated)

PRIMARY OUTCOMES:
Frequency distribution of ABO and Rh blood groups among acute leukemia patients | Between 2022 and 2025
  Assessment of the percentage of each ABO and Rh blood group among patients diagnosed with acute leukemia (including ALL and AML) using retrospectively collected data from blood bank records and clinical files at South Egypt Cancer Institute.

SECONDARY OUTCOMES:
Association between blood group types and leukemia subtype | Between 2022 and 2025
  Evaluation of any statistically significant relationship between specific ABO/Rh blood groups and the type of leukemia (ALL vs AML).

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Mohamed Zahran, M.D., Professor, Principal Investigator — South Egypt Cancer Institute, Assiut University; Walaa Talaat Kamel, M.D., Lecturer, Study Chair — South Egypt Cancer Institute, Assiut University; Esraa Nasr Abd El Hakeem, M.D., Lecturer, Study Chair — Assiut University
Locations (1):
- South Egypt Cancer Institute - Assiut University, Asyut, Egypt

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27069254/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4475644/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/26674825/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7380823/
- See also: Related Info — https://doi.org/10.3389/fmed.2024.1456695
- See also: Related Info — https://www.cancer.org/cancer/leukemia.html